CLINICAL TRIAL: NCT05454436
Title: The Outcome of Healing Intraoral Sinus Tract With a Single or Multi-visit With Bioceramic Sealer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, FAISAL ABDULLAH ALNASSAR, Assistant professor, Department of Restorative Dental Sciences. College of Dentistry,, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1075865046
Record Dates: First submitted 2022-06-15; First posted 2022-07-12 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Sinus Tract; Singler Visit; Multi Visit; Single Cone Obturation Technique; Bioceramic Sealer
MeSH Terms: interventions — Single Person

STUDY DESIGN:
Intervention Model Description: Two group :
  Group A: The treatment will be in a single visit Group B:The treatment will be in Multi visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healing rate of intra oral sinus tract in single visit by SCT with bioceramic sealer (Experimental): When a patient comes with intra oral sinus tract will treat in a single visit. The treatment protocol will be: cleaning and shaping by NITI file ( pro taper gold ) with Naocl 5.25%, EDTA 17% and saline then the canal will be obturate by single cone technique with bioceramic sealer.
  Interventions: Procedure: sinus tract healing in single or multi visit with single cone technique with bioceramic sealer
- Healing rate of intra oral sinus tract in multi visit by SCT with bioceramic sealer (Experimental): When a patient comes with intra-oral sinus tract will treat in a multi-visit. The treatment protocol will : cleaning and shaping by NITI file ( pro taper gold ) with Naocl 5.25%, EDTA 17%, and saline then ca(oh)2 use as Intracanal medication the after disappear the sinus tract the canal will obturate by single cone technique with bioceramic sealer.
  Interventions: Procedure: sinus tract healing in single or multi visit with single cone technique with bioceramic sealer

INTERVENTIONS:
Procedure: sinus tract healing in single or multi visit with single cone technique with bioceramic sealer — Investigators will see the healing rate between single visit and multi visit with single cone technique with bioceramic sealer .

SUMMARY:
The aim of clinical trial is to see is there any difference in the outcome of healing of the intraoral sinus tract when treat in single or multi-visit root canal treatment by an endodontist.

DETAILED DESCRIPTION:
Methods and material :

Inclusion criteria as follows:

Tooth with a sinus tract and radiographic evidence of periradicular bone destruction, Tooth with a necrotic pulp confirmed by pulp tests or with previous root canal treatment, Tooth that was restorable and had an indication for root canal treatment or retreatment, Tooth with a mobility score <3 Absence of periodontal pockets >4 mm deep Patients without significant systemic disease.

Two groups will be divided into:

Group A: will treat in a single visit. The treatment protocol will be: cleaning and shaping by NITI file ( pro taper gold ) with Naocl 5.25%, EDTA 17% and saline then the canal will be obturate by single cone technique with bioceramic sealer.

Group B: will treat in a multi-visit. The treatment protocol will : cleaning and shaping by NITI file ( pro taper gold ) with Naocl 5.25%, EDTA 17% and saline then ca(oh)2 use as Intracanal medication the after disappear the sinus tract the canal will obturate by single cone technique with bioceramic sealer.

Follow-up examinations were performed at 7, 14, and 30 days postoperatively.

According to the clinical, the outcome was classified as:

1. Healed: the sinus tract disappeared completely.
2. Healing: the sinus tract getting smaller and can't be traced with small gutta-percha ( we need to mention GP size)
3. failed: the sinus tract persisted more than 30 days after treatment

ELIGIBILITY:
Inclusion Criteria:

Tooth with a sinus tract and radiographic evidence of periradicular bone destruction, Tooth with a necrotic pulp confirmed by pulp tests or with previous root canal treatment, Tooth that was restorable and had an indication for root canal treatment or retreatment, Tooth with a mobility score <3 Absence of periodontal pockets >4 mm deep Patients without significant systemic disease.

Exclusion Criteria:

Tooth without a sinus tract . Tooth that was not restorable Tooth with a mobility score >3 Absence of periodontal pockets <4 mm deep Patients with significant systemic disease.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — To see is there any significate difference in gender
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Healing rate of intra oral sinus tract in single visit and multi visit root canal treatment | 7 days , 14 days, 30 days
  To see is there sinus tract disappear after treatment

SECONDARY OUTCOMES:
Healing rate of intra oral sinus tract when treat with single cone technique with bioceramic sealer | 7 days , 14 days, 30 days
  Is this technique will effect on healing rate of sinus tract

IPD SHARING:
Plan to Share IPD: Undecided